CLINICAL TRIAL: NCT06214546
Title: Effect of a Body Weight Support System and a Soft Exosuit on Gait in People With Incomplete Spinal Cord Injury
Brief Title: Effect of Different Support Systems on Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Principal Investigator, Noel Keijsers, Prof N.L.W Keijsers, Sint Maartenskliniek
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1124
Record Dates: First submitted 2023-11-23; First posted 2024-01-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: ZeroG; Myosuit; Gait; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Regular walking — Participants perform 6 overground walking trials (12.5 m) without support system. Participants perform all measurements (regular walking, Myosuit, ZeroG) on one single measurement day.
Device: Myosuit — Participants perform 6 overground walking trials (12.5 m) while wearing the Myosuit. ZeroG and Myosuit intervention will be performed in random order.
Device: ZeroG — Participants perform 6 overground walking trials (12.5 m) while walking in the ZeroG. ZeroG and Myosuit intervention will be performed in random order.

SUMMARY:
Body weight support systems are commonly used for gait training. A new breed of devices for gait training are soft exosuits. To optimize rehabilitation outcomes, it is important to gain deeper insight in the effect of these support systems on gait. The aim of this study is to investigate the effect of a body weight support system and soft exosuit on dynamic balance and knee and hip kinematics during gait in people with incomplete spinal cord injury.

DETAILED DESCRIPTION:
Rationale: People with incomplete spinal cord injury (iSCI) often experience gait impairments. Body weight support (BWS) systems are commonly used for gait training. Overground BWS systems could have 2 or 3 degrees of freedom (DoF). A decrease in DoF will reduce the demand's on people's balance capacity during walking. A new breed of devices for gait training are soft exosuits. They could deliver support around the knee and the hip joint, which are the main contributors for bodyweight support. Although a BWS system and a soft exosuit provide both support against gravity these systems differ in the approach of delivering this support. To optimize rehabilitation outcomes, it is important to gain deeper insight in the effect of these support systems on gait. In this study a 2-DoF BWS system, the ZeroG, and a soft exosuit, the Myosuit, will be studied.

Objective: Investigate the effect of a BWS system and soft exosuit on dynamic balance and knee and hip kinematics during gait in people with incomplete spinal cord injury.

Study design: Experimental design.

Study population: Fourteen people with subacute or chronic iSCI (at least 2 weeks after injury) will be included. People with iSCI will be included when having an injury level of C or D on the American Spinal Injury Association Impairment Scale.

Intervention: Participants will visit the Sint Maartenskliniek once and perform overground walking trials in a laboratory setting: regular walking, walking with the ZeroG (BWS system) and walking with the Myosuit (soft exosuit). Each condition consists of 6 walking trials over a distance of 12.5 m.

Main study parameters/endpoints: The main study parameter for dynamic balance during gait will be medio-lateral center of mass excursion. The main study parameter for gait kinematics will be maximum extension of the knee in sagittal plane.

ELIGIBILITY:
Inclusion Criteria:

* People with subacute or chronic iSCI (at least 2 weeks after injury)
* Have an injury level of C or D on the American Spinal Injury Association Impairment Scale
* Age ≥ 18 years
* Walking speed between 0.4 and 0.8 m/s (limited community ambulation) (24)
* Must be able to stand up from a chair without deviating to the left or right side for more than 45 degrees during the movement
* Can walk for 10 meter without the assistance of another person but can be assisted by assistive devices such as, crutches, walking sticks or ankle foot orthoses except knee orthoses or walkers
* Reduced knee and/or hip strength (MRC=<4).

Exclusion Criteria:

* Have another (neurological) disease which can influence motor performance.
* Have wounds
* Taller than 195 and smaller than 150 cm
* Body weight of more than 110 kg or less than 45 kg
* Pregnancy
* Flexion contracture in knee or hip in excess of 10 degrees
* Knee varus malposition in excess of 10 degrees or knee valgus malposition in excess of 10 degrees
* Insufficient mastery of the Dutch language
* Psychiatric backgrounds
* Oncological spinal cord injury
* Stoma
* Unsuitable for participation according to the rehabilitation physician or researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Dynamic balance during gait: medio-lateral center of mass excursion (cm) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Medio-lateral center of mass excursion
Gait kinematics: maximum knee extention | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Maximum extension of the knee in sagittal plane

SECONDARY OUTCOMES:
Dynamic balance during gait: step width (cm) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG.
Gait kinematics: maximum hip extension | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Maximum extension of the hip in sagittal plane
Gait kinematics: range of motion of the knee | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Range of motion of the knee in sagittal plane
Gait kinematics: range of motion of the hip | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Range of motion of the hip in sagittal plane
Gait kinematics: trunk inclination angle | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG. Trunk inclination angle excursion
Walking speed (m/s) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG
Stride length (m) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG
Step time (s) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the Zero.
Double support phase (%) | At baseline (during regular walking, during walking with the Myosuit, during walking with the ZeroG)
  Difference between regular walking, walking with the Myosuit and walking with the ZeroG

OTHER OUTCOMES:
Sex (man/woman) | Subject enrollment
  Descriptive outcome measure
Age (years) | Subject enrollment
  Descriptive outcome measure
Body Mass Index | Subject enrollment
  Descriptive outcome measure. Calculated with weight and height.
Time since spinal cord injury (years) | Subject enrollment
  Descriptive outcome measure.
Spinal cord injury classification defined by the American Spinal Injury Association (ASIA) impairment scale (C or D) | Subject enrollment
  Descriptive outcome measure. The scale has five classification levels (A-E), ranging from complete loss of neural function (A) in the affected area to completely normal (E).
Level of spinal cord injury | Subject enrollment
  Descriptive outcome measure. There are four sections that impact the level of spinal cord injury: cervical, thoracic, lumbar and sacral.

CONTACTS AND LOCATIONS:
Overall Officials: Bart van den Bemt, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No